CLINICAL TRIAL: NCT03193125
Title: Effects of Carnitine Supplementation on Liver Mitochondria Fatty Acid Processing
Brief Title: Carnitine and Liver Mitochondria Fatty Acid Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: University of Tennessee (Other); Touro University (Other)
Responsible Party: Principal Investigator, Owen Carmichael, Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PBRC 2016-076
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Obesity | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carnitine (Experimental): 500 mg of L-carnitine to be taken 3 times a day 15 minutes before meals for 14 days.
  Interventions: Dietary Supplement: L-Carnitine
- Placebo (Placebo Comparator): 500 mg of placebo to be taken 3 times a day 15 minutes before meals for 14 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Carnitine — 500 mg tablets of L-Carnitine taken 3 times daily before meals.
  Arms: Carnitine
Dietary Supplement: Placebo — 500 mg tablets of L-Carnitine taken 3 times daily before meals.
  Arms: Placebo

SUMMARY:
This double-blind, placebo-controlled randomized trial will assess whether 14 days of oral carnitine supplementation modifies mitochondrial fatty acid processing in healthy young adults.

DETAILED DESCRIPTION:
This project will use stable isotope techniques and magnetic resonance spectroscopy (MRS) to take a first step toward clarifying how the benefit of oral carnitine supplementation depends on basal mitochondrial fatty acid processing (MFAP) and MFAP modification, with a specific focus on the liver. Approximately 24 healthy young individuals will be enrolled, with 20 expected to complete. Before and after 14 days of oral carnitine supplementation or placebo, MFAP will be measured using measures of acetyl-carnitine concentration (from long-TE proton MRS) and de novo lipogenesis (DNL, from analysis of blood metabolites following 13C-labeled acetate infusion and high-fructose drink challenge). The MFAP measures will be collected before and after loading participants with a high-fructose drink. Fructose is solely metabolized by the liver.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years
* BMI of 24.5-35.5 kg/m2
* Willingness to eat a prescribed diet of standard meals for a total of six days
* Willingness to undergo carnitine or placebo supplementation for two weeks
* Willingness to undergo study procedures including blood draws, MRS, C13 acetate infusion, DXA, muscle biopsy, and consumption of a sugary drink over the course of 6 hours

Exclusion Criteria:

* Unstable weight in the last 3 months (gain or loss >7 lb (3.2 kg)
* Significant changes in the diet or level of physical activity within the past month
* Clinical history of diabetes or cancer
* Clinically diagnosed heart, kidney, lung, thyroid, liver disease or abnormal liver enzymes that are, in the opinion of the investigator, clinically significant and represent a problem for study inclusion
* Screening fasting glucose > 125 mg/dL
* Screening blood pressure >140 systolic or >90 diastolic
* Use of certain prescribed medications at the discretion of the MI
* Smoking or use of tobacco products in the last 6 months
* Pregnancy or breastfeeding
* Clinically diagnosed neuropsychiatric conditions
* Diets that deviate extremely from the typical western diet in terms of increased meat intake are excluded, at the discretion of the MI.
* Known aversion to or refusal to drink sugary beverages
* Taking any over the counter drugs that alter the intestinal tract, at the discretion of the MI (for example, anti-cholinergic drugs and erythromycin)
* Have taken carnitine supplements regularly in the past 3 months
* Unwilling to discontinue use of dietary supplements containing significant amounts of carnitine or abstain from use one week prior to trial, at the discretion of the MI
* Women who have undergone partial hysterectomy with intact ovarian function
* Standard contra-indications to MRS, including non-removable metallic or electronic implants, claustrophobia or other fear of confinement, or inability to tolerate loud scanner noise
* Calf does not fit into the MRI coil, at the discretion of the PI
* Refusal to allow use of anonymized versions of collected data for research after this study is over

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Liver mitochondrial fatty acid processing | Day 18
  Change from baseline in liver mitochondrial fatty acid processing during high-fructose drink challenge

CONTACTS AND LOCATIONS:
Overall Officials: Owen Carmichael, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized blood assay results, MRI data, and other de-identified clinical lab data will be shared with other researchers beginning 6 months after study completion. It may be obtained through a written request to the PI.